CLINICAL TRIAL: NCT01171170
Title: A Randomized Phase II Study of Paclitaxel-carboplatin-bevacizumab With or Without Nitroglycerin Patches in Patients With Stage IV Non-squamous-non-small Cell Lung Cancer: NVALT12
Brief Title: Paclitaxel-Carboplatin-Bevacizumab +/- Nitroglycerin in Metastatic Non-Squamous-Non-Small Cell Lung Cancer
Acronym: NVALT12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVALT12
Record Dates: First submitted 2010-07-23; First posted 2010-07-28 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; stage IV; nitroglycerin; carboplatin; paclitaxel; bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Bevacizumab; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- carboplatin-paclitaxel-bevacizumab (Active Comparator): paclitaxel 200 mg/m2 d1 - carboplatin area under the curve (AUC) 6 d1 - bevacizumab 15 mg/kg d1. Cycles every 3 weeks. Paclitaxel and carboplatin 4 cycles. Bevacizumab till progression
  Interventions: Drug: carboplatin paclitaxel bevacizumab
- standard treatment plus nitroglycerin (Experimental): paclitaxel 200 mg/m2 d1 - carboplatin AUC 6 d1 - bevacizumab 15 mg/kg d1. Cycles every 3 weeks. Paclitaxel and carboplatin 4 cycles. Bevacizumab till progression. Plus nitroglycerin transdermal patches 25 mg per day from day -3 till +2 of First combination cycle till the last bevacizumab monotherapy cycle
  Interventions: Drug: Standard treatment plus nitroglycerin

INTERVENTIONS:
Drug: carboplatin paclitaxel bevacizumab — paclitaxel 200 mg/m2 d1 - carboplatin AUC 6 d1 - bevacizumab 15 mg/kg d1. Cycles every 3 weeks. Paclitaxel and carboplatin 4 cycles. Bevacizumab till progression
  Other Names: Taxol; Avastin
  Arms: carboplatin-paclitaxel-bevacizumab
Drug: Standard treatment plus nitroglycerin — paclitaxel 200 mg/m2 d1 - carboplatin AUC 6 d1 - bevacizumab 15 mg/kg d1. Cycles every 3 weeks. Paclitaxel and carboplatin 4 cycles. Bevacizumab till progression. Plus nitroglycerin transdermal patches 25 mg per day from day -3 till +2 of First combination cycle till the last bevacizumab monotherapy cycle
  Other Names: Taxol; Avastin
  Arms: standard treatment plus nitroglycerin

SUMMARY:
This study is designed to assess the effects of adding nitroglycerin (NTG) patches, delivery 25 mg NTG per 24 h, to the standard first line treatment of metastatic non-squamous non-small cell lung cancer (NSCLC), i.e. 4 cycles of carboplatin-paclitaxel-bevacizumab, followed by bevacizumab alone until disease progression. Tumor hypoxia is a common phenomenon in lung cancer; it is a known poor prognostic marker, related to treatment resistance. Pre-clinical studies have shown that nitric oxide (NO) donating drugs may decrease hypoxia related drug resistance. NTG is a NO donating drug. NTG increases tumor blood flow and thereby augments antitumor drug delivery to the tumor.

A randomized phase II has shown an increase in the response rate from 42% to 72%, when NTG patches (25 mg/day, day -2 to +3) were added to vinorelbine/cisplatin in patients with advanced NSCLC. In addition, the time to progression increased from 185 to 327 days.

The hypothesis of the present study is that adding NTG transdermal patches to bevacizumab containing chemotherapy improves progression free survival, response rate and overall survival in patients with metastatic non-squamous NSCLC.

DETAILED DESCRIPTION:
Standard treatment for non-small cell lung cancer (NSCLC) consists of platinum-containing chemotherapy. It has been shown that the addition of bevacizumab to standard chemotherapy improves progression-free survival (PFS) and overall survival (OS) in patients with non-squamous NSCLC. There is a need for improved PFS and OS and response rates to chemotherapy are only 25-35%.

Tumor hypoxia is a common phenomenon in lung cancer; it is a known poor prognostic marker, related to treatment resistance. Hypoxia Inducible Factor (HIF) -1α is the major factor regulating the response to hypoxia.

HIF directly activates vascular endothelial growth factor (VEGF) and VEGF-receptor. Bevacizumab interacts with this pathway by blocking VEGF.

Pre-clinical studies have shown that nitric oxide (NO) donating drugs may decrease hypoxia related drug resistance. Nitroglycerin (NTG) is a NO donating drug. NTG increases tumor blood flow and thereby augments antitumor drug delivery to the tumor and inhibits HIF-1α.

Interestingly, it has recently been shown in mouse models that the addition of HIF-1α inhibitors to bevacizumab significantly inhibits tumor growth by inducing apoptosis.

A randomized phase II has shown an increase in the response rate from 42% to 72%, when NTG patches (25 mg/day, day -2 to +3) were added to vinorelbine/cisplatin in patients with advanced NSCLC. In addition, the time to progression increased from 185 to 327 days.

The hypothesis of the present study is that adding NTG transdermal patches to bevacizumab containing chemotherapy improves PFS, response rate and OS in patients with metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven stage IV non-squamous NSCLC (according to IASLC staging 7.0)
* No prior chemotherapy or therapy with systemic anti-tumor therapy (e.g., monoclonal antibody therapy) or prior exposure to agents directed at the HER axis (e.g. epidermal growth factor receptor tyrosine kinase inhibitors (EGFR TKI), Herceptin). Prior surgery and/or localized palliative irradiation is permitted provided that the irradiated lesion is not the only measurable lesion. Prior adjuvant chemotherapy > 1 year ago and prior treatment with an EGFR-TKI for patients with an activating EGFR mutation is allowed.
* Age ≥ 18 years.
* ECOG Performance Status of 0 - 2.
* Life expectancy of at least 12 weeks.
* Subjects with at least one uni-dimensional(for RECIST) measurable lesion.
* Adequate bone marrow, liver and renal function.
* Adequate non-hormonal contraception for females of childbearing potential during the study and in the 6 months thereafter.
* Adequate contraception for male participants (or their partners) during the study and in the 6 months thereafter.

Exclusion Criteria:

* Clinically significant (i.e. active) cardiovascular disease: congestive heart failure >NYHA class 2; CVA or myocardial infarction < 6 months prior to study entry; uncontrolled hypertension (blood pressure systolic > 150 mmHg and/or diastolic > 100 mmHg).
* Symptomatic hypotension.
* History of hemoptysis at least grade 2 (bright red blood of at least 2,5 ml in the last 3 months)
* Evidence of tumor invading major blood vessels on imaging (i.e. superior vena cava or pulmonary artery).
* History of HIV infection or chronic hepatitis B or C.
* Active clinically serious infection
* Symptomatic metastatic brain or meningeal tumors. Patients with brain metastasis may be included the patient is treated with brain radiotherapy and asymptomatic.
* History of organ allograft.
* Patients with evidence or history of bleeding diathesis.
* Non-healing wound or ulcer.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry
* Radiotherapy within 4 weeks of start of study drug. Palliative radiotherapy for bone lesions is allowed > 14 days of start of chemotherapy. Major surgery within 4 weeks of start of study.
* Use of vasodilators (including 5-phosphodiesterase inhibitors, calcium antagonists or nitrates)
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
progression free survival | every 6 weeks during chemotherapy
  Imaging

SECONDARY OUTCOMES:
objective response rate | every 6 weeks during chemotherapy
  Imaging
disease control rate | every 6 weeks during chemotherapy
  Imaging
duration of response | every 6 weeks during chemotherapy
  Imaging
safety of the treatment | every 3 weeks during chemotherapy
  adverse events, hematology, chemistry, physial examination
prediction of early response | after 3 weeks
  FDG PET scan (exploratory objective)
decreased hypoxia | after 6 weeks
  FAZA scan (exploratory objective)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie C. Dingemans, MD PhD, Principal Investigator — Maastricht UMC
Locations (8):
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - VU medisch centrum, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Catharina-Ziekenhuis, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Maastricht UMC, Maastricht
  - HagaZiekenhuis, The Hague
  - Isala Klinieken, Zwolle

REFERENCES:
- [Result] Dingemans AM, Groen HJ, Herder GJ, Stigt JA, Smit EF, Bahce I, Burgers JA, van den Borne BE, Biesma B, Vincent A, van der Noort V, Aerts JG; NVALT study group. A randomized phase II study comparing paclitaxel-carboplatin-bevacizumab with or without nitroglycerin patches in patients with stage IV nonsquamous nonsmall-cell lung cancer: NVALT12 (NCT01171170)dagger. Ann Oncol. 2015 Nov;26(11):2286-93. doi: 10.1093/annonc/mdv370. Epub 2015 Sep 7. PMID 26347109
- [Result] de Jong EE, van Elmpt W, Leijenaar RT, Hoekstra OS, Groen HJ, Smit EF, Boellaard R, van der Noort V, Troost EG, Lambin P, Dingemans AC. [18F]FDG PET/CT-based response assessment of stage IV non-small cell lung cancer treated with paclitaxel-carboplatin-bevacizumab with or without nitroglycerin patches. Eur J Nucl Med Mol Imaging. 2017 Jan;44(1):8-16. doi: 10.1007/s00259-016-3498-y. Epub 2016 Sep 6. PMID 27600280
- [Result] Degens JHRJ, Sanders KJC, de Jong EEC, Groen HJM, Smit EF, Aerts JG, Schols AMWJ, Dingemans AC. The prognostic value of early onset, CT derived loss of muscle and adipose tissue during chemotherapy in metastatic non-small cell lung cancer. Lung Cancer. 2019 Jul;133:130-135. doi: 10.1016/j.lungcan.2019.05.021. Epub 2019 May 20. PMID 31200819
- [Result] de Goeje PL, Poncin M, Bezemer K, Kaijen-Lambers MEH, Groen HJM, Smit EF, Dingemans AC, Kunert A, Hendriks RW, Aerts JGJV. Induction of Peripheral Effector CD8 T-cell Proliferation by Combination of Paclitaxel, Carboplatin, and Bevacizumab in Non-small Cell Lung Cancer Patients. Clin Cancer Res. 2019 Apr 1;25(7):2219-2227. doi: 10.1158/1078-0432.CCR-18-2243. Epub 2019 Jan 14. PMID 30642911
- [Derived] de Jong EEC, Hendriks LEL, van Elmpt W, Gietema HA, Hofman PAM, De Ruysscher DKM, Dingemans AC. What you see is (not) what you get: tools for a non-radiologist to evaluate image quality in lung cancer. Lung Cancer. 2018 Sep;123:112-115. doi: 10.1016/j.lungcan.2018.07.014. Epub 2018 Jul 18. PMID 30089580
- See also: Related Info — http://www.nvalt.nl